CLINICAL TRIAL: NCT06818812
Title: A Phase 1, Open-Label, Multicenter Study of INCB186748 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation
Brief Title: A Study to Evaluate INCB186748 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB186748-101; 2024-519018-30-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors
Keywords: INCB186748; KRASG12D Mutation; pancreatic ductal adenocarcinoma (PDAC); colorectal cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1a: Dose Escalation monotherapy (Experimental): INCB186748 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB186748
- Part 1b: Dose Expansion monotherapy (Experimental): INCB186748 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB186748
- Part 1c: Pharmacodynamic cohort (Experimental): INCB186748 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB186748
- Part 1d: Food-Effect (Experimental): Evaluate food effect on drug exposure as defined in the protocol.
  Interventions: Drug: INCB186748
- Part 2a: Dose Escalation combination (Experimental): INCB186748 in combination at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB186748; Drug: Cetuximab; Drug: GEMNabP; Drug: mFOLFIRINOX
- Part 2b: Dose Expansion combination (Experimental): INCB186748 in combination at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB186748; Drug: Cetuximab; Drug: GEMNabP; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: INCB186748 — INCB186748 will be administered at protocol defined dose.
Drug: Cetuximab — Cetuximab will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: GEMNabP — GEMNabP will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: mFOLFIRINOX — mFOLFIRINOX will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination

SUMMARY:
The purpose of this study is to evaluate INCB186748 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Locally advanced or metastatic solid tumor with KRAS G12D mutation.
* For Part 1 and Part 2 Combination Group 1: Disease progression on or after prior standard treatment, or intolerance to or ineligibility for standard treatment, or no standard available treatment to improve the disease outcome.
* For Part 2 Combination Groups 2 and 3: No more than 1 prior standard treatment.
* Cohort-specific requirements as follows:

  * Parts 1a and 1d: histologically or cytologically confirmed malignant solid tumor of any tissue origin.
  * Part 1b

    * Disease Group 1: diagnosis of PDAC and at least 1 but no more than 2 prior standard systemic regimens for pancreatic cancer.
    * Disease Group 2: diagnosis of CRC.
  * Part 1c: Confirmed diagnosis of PDAC or CRC.
  * Parts 2a and 2b

    * Combination Group 1 (INCB186748 in combination with cetuximab):

      * Diagnosis of PDAC or
      * Diagnosis of CRC and ∘ Prior treatment in the advanced setting with a fluoropyrimidine-based chemotherapy regimen containing either oxaliplatin or irinotecan and

        * In Part 2a: ≤ 3 prior standard regimens.
        * In Part 2b: ≤ 2 prior standard regimens.
    * Combination Group 2 (INCB186748 in combination with GEMNabP) and
    * Combination Group 3 (INCB186748 in combination with mFOLFIRINOX):

      * Diagnosis of PDAC.
      * ≤ 1 prior standard systemic regimen for pancreatic cancer.
* Measurable disease according to RECIST v1.1.
* ECOG performance status score of 0 or 1.

Exclusion Criteria:

* Prior treatment with any KRAS inhibitor.
* Known additional invasive malignancy within 1 year of the first dose of study drug.
* History of organ transplant, including allogeneic stem cell transplantation.
* Significant, uncontrolled medical condition.
* History or presence of an ECG abnormality.
* Inadequate organ function.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-03-27 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 12 months and 60 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event occurring after the first dose of study drug up to 30 days (for INCB186748 as monotherapy and in combination with GEMNabP or mFOLFIRINOX) and 60 days (for INCB186748 in combination with cetuximab) after the last dose of INCB186748.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to approximately 12 months and 60 days
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
INCB186748 pharmacokinetic (PK) in Plasma | Up to approximately 12 months
  INCB186748 concentration in plasma.
Objective Response Rate (ORR) | Up to approximately 12 months
  Defined as having a best overall Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Disease Control Response (DCR) | Up to approximately 12 months
  Defined as having a best overall response of CR, PR, or Stable Disease (SD) as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Duration of Response (DOR) | Up to approximately 12 months
  Defined as the time from earliest date of disease response (Completed Response or Partial Response) until earliest date of disease progression as determined by the investigator by radiographic disease assessment according to RECIST v1.1 or death due to any cause if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (9):
- United States (9):
  - UCLA Healthcare Hematology-Oncology, Santa Monica, California
  - Sarah Cannon Research Institue At Healthone, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Sarasota, Florida
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Scri Oncology Partners, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate INCB186748 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation — https://www.incyteclinicaltrials.com/study/?id=INCB186748-101&SearchTerm=INCB186748-101&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=